CLINICAL TRIAL: NCT00599404
Title: An Open-Label, 2-Period Pharmacokinetic Study to Evaluate the Intra-Subject Variability in Esomeprazole Plasma Levels in Healthy Subjects Following Oral Administration of PN 400 Tablets
Brief Title: PK Study to Evaluate Esomeprazole Plasma Levels Following Administration of PN 400
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: POZEN (Industry)
Responsible Party: David Taylor, Pozen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PN400-111
Record Dates: First submitted 2008-01-11; First posted 2008-01-23 (Estimated); Last update posted 2008-04-30 (Estimated); Status verified 2008-04

CONDITIONS: Healthy
Keywords: Pharmacokinetics study

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: PN400 — 500 mg esomeprazole/20 mg naproxen, once daily on Days 1-10 and twice daily on Days 2-9

SUMMARY:
Pharmacokinetic study in healthy subjects with single and repeat b.i.d. dosing of PN 400 tablets from the same drug product batch.

ELIGIBILITY:
Inclusion Criteria:

Healthy male or non-pregnant female subjects between 18-55 years of age as well as other standard inclusion criteria for a study of this nature

Exclusion Criteria:

Standard inclusion criteria for a study of this nature

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2008-01; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic profile following dosing with PN400 | 24-hour PK on Day 1 & Day 10 of each treatment period

SECONDARY OUTCOMES:
To evaluate the safety of PN400 | Day 1-10 of each treatment period